CLINICAL TRIAL: NCT04201613
Title: Robot-Enhanced Stroke Therapy Optimized Rehabilitation
Brief Title: Robot-Enhanced Stroke Therapy Optimizes Rehabilitation (RESTORE)
Acronym: RESTORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Sean Dukelow, Associate Professor of Physical Medicine and Rehabilitation, University of Calgary
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: REB13-0414
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Stroke
Keywords: Stroke; Stroke Rehabilitation; Robotic Exoskeleton
MeSH Terms: conditions — Stroke | interventions — Exoskeleton Device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Early Robotic Rehab Low Intensity (Active Comparator): This group will begin robotic rehabilitation using a robotic exoskeleton between days 5-9 after their stroke. They will receive one hour of treatment per day for 20 days.
  Interventions: Device: Robotic exoskeleton
- Early Robotic Rehab High Intensity (Active Comparator): This group will begin robotic rehabilitation using a robotic exoskeleton between days 5-9 after their stroke. They will receive 2 one-hour treatment sessions per day for 20 days.
  Interventions: Device: Robotic exoskeleton
- Late Robotic Rehab Low Intensity (Active Comparator): This group will begin robotic rehabilitation using a robotic exoskeleton between days 21-25 after their stroke. They will receive one hour of treatment per day for 20 days.
  Interventions: Device: Robotic exoskeleton
- Late Robotic Rehab High Intensity (Active Comparator): This group will begin robotic rehabilitation using a robotic exoskeleton between days 21-25 after their stroke. They will receive 2 one-hour treatment sessions per day for 20 days.
  Interventions: Device: Robotic exoskeleton
- Control Group (Active Comparator): This group will receive usual care with robotic assessment.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Device: Robotic exoskeleton — The Kinesiological Instrument for Normal and Altered Reaching Movements (KINARM) robotic exoskeleton used to provide therapy and assessment. The device has framework that supports the arms and the supports are adjustable to ensure a comfortable fit. Motors attached to the framework record shoulder and elbow movements and also move the arms.
  Other Names: KINARM
  Arms: Early Robotic Rehab High Intensity; Early Robotic Rehab Low Intensity; Late Robotic Rehab High Intensity; Late Robotic Rehab Low Intensity
Behavioral: Usual Care — This group will receive standard care with no additional therapy.
  Arms: Control Group

SUMMARY:
The purpose of this study is to investigate two aspects of robotic therapy after stroke. One goal is to determine if early robotic rehabilitation of the upper limb (beginning 5-9 days post-stroke) is more effective than later robotic rehabilitation (beginning 21-25 days post-stroke). The other goal is to determine if higher intensity robotic rehabilitation (2 hours/day) is more effective than lower intensity robotic rehabilitation (1 hour/day).

DETAILED DESCRIPTION:
Medically stable stroke subjects will be recruited in the first few days following their stroke. All participants will complete clinical and robotic assessments of neurologic function at 7 time points. Therapy will occur daily (Monday through Friday) for 20 days.

Study participants will be randomly assigned to 1) start robot therapy early or late after stroke and 2)receive one or two hours of robot therapy per treatment day for four weeks, or 3) control group that will receive the current standard of care.

The participant's chart will be reviewed for information about their stroke and related health effects and medical treatments. Assessment points to track progress will occur at 7, 18, 31,44,90,180, and 365 days after a stroke for all groups (give or take 2 days to account for weekends and holidays).

Standard clinical assessments of neurologic function will be done at each assessment point and include: cognition, arm strength, muscle tone, spasticity, reflexes, dexterity, visual acuity and fields, the Behavioural Inattention Test, and tests of arm movement (Fugl-Meyer Upper-Extremity, Box and Block Test, Chedoke-McMaster Stroke Assessment, and the Action Research Arm Test). These assessments can usually be done in about an hour. The assessment may be done over two sessions if needed due to fatigue or scheduling conflicts.

Robotic therapy will be conducted using the Kinesiological Instrument for Normal and Altered Reaching Movements (KINARM, Bkin Technologies, Kingston, ON). It will include several different tasks, each designed to train aspects of sensorimotor function of the proximal upper limb. Task performance will be monitored and difficulty will increase within and between sessions. The majority of the investigator's methods have been used previously to achieve equivalent or superior outcomes to standard rehabilitation.

Robotic assessment will measure elbow and shoulder range of motion, reaching for targets, the ability to mirror match the position of an arm with the other arm, and the ability to use both arms to hit away moving targets. The robotic assessment will take approximately 1.5 hours.

Robotic tasks include:

Visually guided reaching with assistance or resistance; Virtual Soccer; Shape Tracking; Whack-a-mole; Table Tennis Task; Ball on Bar Task; Proprioceptive Reaching; Hand Ball; Proprioceptive Shape Tracking.

ELIGIBILITY:
Inclusion Criteria:

* Recent first stroke (ischemic or hemorrhagic)
* Upper extremity Fugl-Meyer score 15-45
* Modified Ashworth score of shoulder/elbow less than or equal to 2
* Able to follow task instructions
* Visual acuity better than 20/50 in both eyes
* Able to give consent
* Able to commit to follow-up

Exclusion Criteria:

* Prior stroke or significant neurologic problem (e.g. Multiple Sclerosis)
* Pre-existing musculoskeletal injury that will interfere with active therapy
* Pre-Stroke Modified Rankin Score > 2
* Clinical evidence of Unilateral Spatial Neglect on the Behavioural Inattention Test (BIT)
* Enrollment in a concurrent clinical intervention trial
* Major co-morbid or concurrent illness such that improvement is unlikely or completion of the protocol as specified is unlikely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer upper extremity motor function score (FMA) | From baseline to 44 days
  FMA scores upper extremity motor impairment based on 22 items and scores range from 0 (completely plegic) to 66 (normal).

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | From baseline to 180 days
  FIM rates subjects on 18 items across many functions such as eating, grooming, bathing and dressing on a scale from 1 (total assistance needed) to 7 (complete independence). Lowest possible score is 18 (lowest independence) and the best possible score is 126 (completely independent). The FIM is the standard measure used by rehabilitation facilities in Cananda and the United States to evaluate overall function and burden of care.
modified Rankin Scale (mRS) | From baseline to 180 days
  The mRS is a disability rating scale from 0 (no symptoms at all) to 6 (deceased).
Action Research Arm Test (ARAT) | From baseline to 180 days
  The ARAT assesses arm function to determine the quality of the arm movement, and the limitation of activity. The ARAT consists of 4 sub-tests; that examines and individual's grip, grasp, pinch and gross motor movement in order to determine upper extremity function. Objects of varying size, shape, and weight must be either grasped, handled or moved in a specific task in order to evaluate function. Low scores mean worse function with the minimum possible score being 0 and the highest possible score being 57 (normal function).
Robotic Assessments | From baseline to 180 days.
  Robotic Assessments. The robotic assessment consists of a number of upper limb tests of neurologic function which have been validated against standard clinical measures. Tasks include: Range of Motion, Visually Guided Reaching, Limb Position Matching, Limb Kinesthesia, and Object Hit. These assessments use z-scores, based on normal distributions, as a measure of performance. Scores within 1.96 standard deviations away from 0 are considered normal and scores beyond 1.96 standard deviations are considered impaired.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Dukelow, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Volpe BT, Krebs HI, Hogan N, Edelstein OTR L, Diels C, Aisen M. A novel approach to stroke rehabilitation: robot-aided sensorimotor stimulation. Neurology. 2000 May 23;54(10):1938-44. doi: 10.1212/wnl.54.10.1938. PMID 10822433
- [Background] Fasoli SE, Krebs HI, Stein J, Frontera WR, Hogan N. Effects of robotic therapy on motor impairment and recovery in chronic stroke. Arch Phys Med Rehabil. 2003 Apr;84(4):477-82. doi: 10.1053/apmr.2003.50110. PMID 12690583
- [Background] Dukelow SP, Herter TM, Moore KD, Demers MJ, Glasgow JI, Bagg SD, Norman KE, Scott SH. Quantitative assessment of limb position sense following stroke. Neurorehabil Neural Repair. 2010 Feb;24(2):178-87. doi: 10.1177/1545968309345267. Epub 2009 Sep 30. PMID 19794134
- [Background] Ferraro M, Palazzolo JJ, Krol J, Krebs HI, Hogan N, Volpe BT. Robot-aided sensorimotor arm training improves outcome in patients with chronic stroke. Neurology. 2003 Dec 9;61(11):1604-7. doi: 10.1212/01.wnl.0000095963.00970.68. PMID 14663051
- [Background] Daly JJ, Hogan N, Perepezko EM, Krebs HI, Rogers JM, Goyal KS, Dohring ME, Fredrickson E, Nethery J, Ruff RL. Response to upper-limb robotics and functional neuromuscular stimulation following stroke. J Rehabil Res Dev. 2005 Nov-Dec;42(6):723-36. doi: 10.1682/jrrd.2005.02.0048. PMID 16680610
- [Background] Finley MA, Fasoli SE, Dipietro L, Ohlhoff J, Macclellan L, Meister C, Whitall J, Macko R, Bever CT Jr, Krebs HI, Hogan N. Short-duration robotic therapy in stroke patients with severe upper-limb motor impairment. J Rehabil Res Dev. 2005 Sep-Oct;42(5):683-92. doi: 10.1682/jrrd.2004.12.0153. PMID 16586194
- [Background] Volpe BT, Lynch D, Rykman-Berland A, Ferraro M, Galgano M, Hogan N, Krebs HI. Intensive sensorimotor arm training mediated by therapist or robot improves hemiparesis in patients with chronic stroke. Neurorehabil Neural Repair. 2008 May-Jun;22(3):305-10. doi: 10.1177/1545968307311102. Epub 2008 Jan 9. PMID 18184932
- [Background] Lo AC, Guarino PD, Richards LG, Haselkorn JK, Wittenberg GF, Federman DG, Ringer RJ, Wagner TH, Krebs HI, Volpe BT, Bever CT Jr, Bravata DM, Duncan PW, Corn BH, Maffucci AD, Nadeau SE, Conroy SS, Powell JM, Huang GD, Peduzzi P. Robot-assisted therapy for long-term upper-limb impairment after stroke. N Engl J Med. 2010 May 13;362(19):1772-83. doi: 10.1056/NEJMoa0911341. Epub 2010 Apr 16. PMID 20400552
- [Background] Liao WW, Wu CY, Hsieh YW, Lin KC, Chang WY. Effects of robot-assisted upper limb rehabilitation on daily function and real-world arm activity in patients with chronic stroke: a randomized controlled trial. Clin Rehabil. 2012 Feb;26(2):111-20. doi: 10.1177/0269215511416383. Epub 2011 Aug 12. PMID 21840917
- [Background] Cumming TB, Thrift AG, Collier JM, Churilov L, Dewey HM, Donnan GA, Bernhardt J. Very early mobilization after stroke fast-tracks return to walking: further results from the phase II AVERT randomized controlled trial. Stroke. 2011 Jan;42(1):153-8. doi: 10.1161/STROKEAHA.110.594598. Epub 2010 Dec 9. PMID 21148439
- [Background] Hu MH, Hsu SS, Yip PK, Jeng JS, Wang YH. Early and intensive rehabilitation predicts good functional outcomes in patients admitted to the stroke intensive care unit. Disabil Rehabil. 2010;32(15):1251-9. doi: 10.3109/09638280903464448. PMID 20131942
- [Background] Scott SH, Dukelow SP. Potential of robots as next-generation technology for clinical assessment of neurological disorders and upper-limb therapy. J Rehabil Res Dev. 2011;48(4):335-53. doi: 10.1682/jrrd.2010.04.0057. PMID 21674387
- [Background] Semrau JA, Herter TM, Scott SH, Dukelow SP. Robotic identification of kinesthetic deficits after stroke. Stroke. 2013 Dec;44(12):3414-21. doi: 10.1161/STROKEAHA.113.002058. Epub 2013 Nov 5. PMID 24193800
- [Derived] Keeling AB, Piitz M, Semrau JA, Hill MD, Scott SH, Dukelow SP. Robot enhanced stroke therapy optimizes rehabilitation (RESTORE): a pilot study. J Neuroeng Rehabil. 2021 Jan 21;18(1):10. doi: 10.1186/s12984-021-00804-8. PMID 33478563